CLINICAL TRIAL: NCT00200941
Title: A Randomized, Double-Blind, Placebo-Controlled, Parallel Group Study to Determine the Effacy and Safety of Topiramate in Subjects With Restless Legs Syndrome (RLS)
Brief Title: Efficacy and Safety Study of Topiramate to Treat Restless Legs Syndrome
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Neurocare (Other)
Collaborators: Ortho-McNeil Pharmaceutical (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Educational/Counseling/Training
Other Study IDs: CAPSS-178
Record Dates: First submitted 2005-09-12; First posted 2005-09-20 (Estimated); Last update posted 2005-12-16 (Estimated); Status verified 2005-09

CONDITIONS: Restless Legs Syndrome
Keywords: Restless Legs Syndrome; Topiramate; Actigraphy; Polysomnography
MeSH Terms: conditions — Restless Legs Syndrome | interventions — Topiramate

INTERVENTIONS:
Drug: Topiramate

SUMMARY:
This study is intended to determine whether topiramate is an efficacious and safe treatment for restless legs syndrome.

DETAILED DESCRIPTION:
Benzodiazepines, levo-dopa/carbidopa, dopamine agonists, anticonvulsants, and opioids have been used with variable success, to treat RLS. Often, RLS patients treated with a benzodiazepine, over the course of several months, develop tolerance to the medication. Also, benzodiazepines can cause confusion or daytime sleepiness and may be addictive. Patients may also develop tolerance to levo-dopa/carbidopa treatment. Because of the short half-life, symptoms may be suppressed for only the first part of the sleep period and then recur later during the night. Rebound has been reported. Worse yet, augmentation, the occurrence of RLS symptoms, often more severe than before treatment began, earlier in the day, may occur in up to 80% of RLS patients treated with levod-dopa/carbidopa. Dopamine agonists, including pergolide, pramipexole, and ropinirole, are effective for some patients but not for others. Common side effects of these drugs include coryza, hypotension, and rash. Of the anticonvulsants, preliminary reports suggest that gabapentin, carbamazepine, and divalproex can suppress RLS symptoms in some patients, especially those with mild RLS. Side effects include sleepiness, ataxia, and weight gain. Opioid treatment for RLS has been described as effective but, aside from the stigma of taking controlled substances regularly, side effects may include nausea, sedation, constipation, and dysequilibrium. Iron supplementation is therapeutic in some patients with iron deficiency and RLS.

Preliminary anecdotal data suggest that topiramate reduces RLS symptoms. Topiramate has several potential mechanisms of action including enhancement of GABA-mediated inhibition, which may account for the observed benefit in patients with RLS.

Topiramate may be a better alternative than the currently available treatments to suppress RLS symptoms. Like gabapentin, it offers the possibility of decreasing RLS symptoms while also diminishing pain, especially in those patients who have limb pain from neuropathy, radiculopathy, or other causes. Unlike gabapentin, topiramate may help overweight patients with RLS lose weight, if anedotal reports on weight reduction with the medication are correct.

ELIGIBILITY:
Inclusion Criteria:

* The symptoms of each subject must meet the diagnostic criteria of the International RLS Study Group
* More than five periodic leg movements per hour recorded during baseline polysomnography (PSG)
* Each subject must discontinue all treatments for RLS and agreed not to take other RLS treatments during the study

Exclusion Criteria:

* Clinically unstable medical problems
* History of nephrolithiasis
* Progressive neurologic disease
* Inadequate therapeutic response from two previous treatment regimens for RLS
* Subjects unable to discontinue medications known to cause or suppress RLS
* Subjects with sleep apnea syndrome
* Subjects consuming daily more than three beverages containing caffeine

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 44
Dates: Start 2001-08; Study Completion 2005-04

PRIMARY OUTCOMES:
The average number of periodic leg movements during three consecutive nights of actigraphy beginning at the end of the double blind phase

SECONDARY OUTCOMES:
Proportion of time in bed without leg movements during the three consecutive nights of actigraphy beginning at the end of the double blind phase
SF-36 at the last visit of the double blind phase
Score on the RLS Rating Scale (modified) questionnaire at the last visit of the double blind phase
Periodic leg movements during sleep and wakefulness during the PSG recorded at the end of the double blind phase
PSG measures including periodic leg movement arousal index, latency until sustained sleep, sleep efficacy, and wake after sleep onset
Sleep diaries at the last double-blind visit
Epworth sleepiness scale at the last double-blind visit

CONTACTS AND LOCATIONS:
Overall Officials: Michael P Biber, MD, Principal Investigator — Neurocare
Locations (1):
- Neurocare, Newton, Massachusetts, United States